CLINICAL TRIAL: NCT03148535
Title: Clinical Psychopharmacology Division Institute of Mental Health, Peking University
Brief Title: Guidance Model of Standardized Treatment of Antidepressants in Bipolar Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Si Tianmei, Clinical Psychopharmacology Division Institute of Mental Health, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1-4111
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: the Use of Antidepressants in Patients With Bipolar Depression
MeSH Terms: interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lithium carbonate (Experimental): recieve lithium carbonate
  Interventions: Drug: Lithium Carbonate
- lithium carbonate combined with SSRI antidepressant treatment (Experimental): recieve lithium carbonate combined with SSRI antidepressant treatment
  Interventions: Drug: lithium carbonate combined with SSRI antidepressant treatment

INTERVENTIONS:
Drug: Lithium Carbonate — bipolar depression recieve lithium Carbonate treatment
  Arms: lithium carbonate
Drug: lithium carbonate combined with SSRI antidepressant treatment — lithium carbonate combined with SSRI antidepressant treatment
  Arms: lithium carbonate combined with SSRI antidepressant treatment

SUMMARY:
The bipolar depression patients of 18-55 years old were recruited. At the time of enrollment, the demographic, symptomatic, neuropsychological, neurobiological and genetic data was collected. After the completion of the baseline assessment and examination, the patients were given lithium carbonate or lithium carbonate combined with SSRI antidepressant treatment. Clinical evaluation was performed at 2 and 8 weeks after treatment, including the therapeutic efficacy and adverse drug reactions, and monitoring of serum lithium concentration. The patients further receive the fMRI scans after treatment for 8 weeks. Through above work, this study aimed to provide some guidance for the use of antidepressants in patients with bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* age 18-55 years old, bipolar depression

Exclusion Criteria:

* other mental illness, serious somatic illnesses, MRI contradictions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
HRSD reduction ratio | 8 weeks
  HRSD reduction ratio

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Institute of mental health, Peking University, Beijing, Beijing Municipality
  - The first hospital of Hebei Province University, Shijiazhuang, Hebei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Dalian No.7 People's Hospital, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: No